CLINICAL TRIAL: NCT03387007
Title: Effect of Psycho-social Support Training by School Teachers on Improving Mental Health and Hope of School Going Adolescents in Earthquake Affected Districts in Nepal
Brief Title: Psycho-social Support on Mental Health and Hope of Adolescents Affected by Earthquake in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Rolina Dhital, PhD Candidate, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUniversity
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse)
Keywords: adolescent; mental health; hope; psycho-social support; school teachers; earthquake
MeSH Terms: conditions — Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Two teachers from each of the schools included in this arm received training on providing psycho-social support to their students to be implemented in their regular routine school activities
  Interventions: Behavioral: Psychosocial support training for school teachers
- Control (No Intervention): The teachers from the schools in this arm did not receive training on psycho-social support

INTERVENTIONS:
Behavioral: Psychosocial support training for school teachers — The intervention for this study was schoolteachers' training on psychosocial support.A clinical psychologist provided 2-day training (a total of 16 hours) training on psychosocial support for the schoolteachers
  Arms: Intervention

SUMMARY:
Adolescents are prone to mental health problems such as post-traumatic stress disorder (PTSD) and depression which could become worse in the aftermath of disasters. However, hope can help adolescents cope with the challenges better. For resource poor disaster prone settings, school teachers can provide timely psycho-social support that could improve mental health and hope among adolescents.

Nepal is a disaster prone country that faced a devastating earthquake in 2015 that claimed thousands of lives and left many homeless which could have affected the mental health of adolescents.This study was conducted in schools of Dhading, a severely earthquake affected district and schools of Myagdi, a least affected district by earthquake in Nepal. The intervention focused on training school teachers on psycho-social support for adolescents.

DETAILED DESCRIPTION:
Adolescents are prone to mental health problems such as post-traumatic stress disorder (PTSD) and depression which could become worse in the aftermath of disasters. However, some adolescents can have better hope that helps them to cope with the challenges following adverse events such as earthquake.

Nepal is a low income and disaster prone country that ranks 11th for earthquake risks globally. In April 2015, the country faced a devastating earthquake of 7.8 Magnitude that killed thousands of people. Fourteen out of seventy five districts in Nepal were declared as severely affected districts.

However, the adolescents may not have received enough psychosocial support after the earthquake. The damage caused by earthquake was further worsened by the political instability in the country leading to delay in reconstruction work in earthquake-affected areas. Difficult circumstances following the earthquake could have affected the mental of adolescents negatively. However, the evidence on mental health status of adolescents following massive disaster such as earthquake remains inadequate.

For resource poor and disaster prone settings such as Nepal, school teachers can provide timely psychosocial support that could improve mental health and hope among adolescents. School based teacher mediated interventions could be more sustainable and feasible in the complex scenario of post-disaster settings. However, evidence on teacher mediated interventions in low resource disaster settings remain inadequate.

The objectives of this study were to assess mental health and level of hope among the adolescents in selected districts and examine the effect of school teachers' training on psychosocial support on mental health and hope among the adolescents.

The intervention for this study was schoolteachers' training on psycho-social support. A clinical psychologist provided 2-day training on psycho-social support for 22 schoolteachers (2 teachers from each intervention school). The training guidelines were adapted from the United Nations Relief and Works Agency (UNRWA) on psycho-social support for education in emergencies. The training provided basic skills to the schoolteachers so that they will be able to provide psycho-social support for children affected. The lesson learned from the training was intended to be applied by the school teachers in their everyday regular school activities. A follow up study was conducted at 6 months follow up among the adolescents to assess the change in their mental health status and hope.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents studying in grade 6, 7 and 8 of the selected schools at the time of data collection
* Adolescents with written consent from themselves and their guardian

Exclusion Criteria:

* Adolescent who refused to participate

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1912 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline post traumatic stress symptoms at 6 months | baseline and 6 month follow up
  Post traumatic stress disorder symptoms among adolescents using Child post traumatic symptom scale symptom scale which is a 17 item scale. The minimum score is 0 and maximum score is 52. Higher score indicates higher symptoms for PTSD.
Change from baseline depression symptoms at 6 months | baseline and 6 month follow up
  Depression symptoms among adolescents using depression self rating scale which is an 18 item scale. The minimum score is 0 and maximum score is 36. Higher scores indicate higher symptoms for depression.
Change from baseline hope at 6 months | baseline and 6 month follow up
  Hope as an antecedent of resilience and positive aspect of mental health using Children's Hope scale which is a 6 item scale. The minimum score is 0 and maximum score is 1 and maximum score is 36. The higher score indicate higher hope.

CONTACTS AND LOCATIONS:
Overall Officials: Rolina Dhital, MHSc, Principal Investigator — Tokyo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhital R, Shibanuma A, Miyaguchi M, Kiriya J, Jimba M. Effect of psycho-social support by teachers on improving mental health and hope of adolescents in an earthquake-affected district in Nepal: A cluster randomized controlled trial. PLoS One. 2019 Oct 1;14(10):e0223046. doi: 10.1371/journal.pone.0223046. eCollection 2019. PMID 31574127